CLINICAL TRIAL: NCT05515926
Title: Physiological Responses to Osteopathic Manipulative Techniques in Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Touro University Nevada (Other)
Responsible Party: Principal Investigator, Marina Ioudina, Assistant Professor, Touro University Nevada
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TUN IRB4-10-13A
Record Dates: First submitted 2022-07-27; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Healthy Young Adults
Keywords: Osteopathic manipulation; Autonomic; Cardiovascular
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cranial OMT (Experimental): The experimental group received the three cranial osteopathic manipulative techniques, occipital-atlantal decompression (OAD), occipital-mastoid decompression (OMD), and compression of the fourth ventricle (CV4), consecutively applied.
  Interventions: Procedure: Cranial manipulation group, or cranial osteopathic techniques (OMM)
- Sham manipulation (Sham Comparator): The osteopathic physician placed his hands on the skull of the subject but did not influence cranial motion.
  Interventions: Procedure: Sham manipulation
- Non touch group (No Intervention): The control group whose members did not receive any manipulations.

INTERVENTIONS:
Procedure: Cranial manipulation group, or cranial osteopathic techniques (OMM) — Cranial OMT procedure:
  Subjects were relaxed and lying on the back for entire time of the research protocol (approximately 30 min). Osteopathic physician performed the osteopathic manipulations using his hands. The physician gently applied a small amount of force to the neck and head to release tissue tension until feeling a softening and warmth of tissues. Subjects experienced a sensation of slight pulling, releasing, or relaxing of the tissue.
  Other Names: Cranial osteopathic manipulations, cranial osteopathic techniques, cranial OMT procedure
  Arms: Cranial OMT
Procedure: Sham manipulation — The osteopathic physician placed his hands on the skull of the subject but did not influence cranial motion.
  Other Names: Sham
  Arms: Sham manipulation

SUMMARY:
This study was designed to investigate the effect of selected osteopathic manipulative techniques (OMT) on cardiovascular functions in healthy young men and women.

This work addressed questions regarding physiological responses to OMT in maintaining the cardiovascular homeostasis by (1) measuring changes in the cardiac autonomic nerves activity, (2) measuring changes in cardiovascular parameters such as blood pressure, cardiac contractility, and heart rate, and (3) investigating if changes in the cardiac autonomic nerves activity were related to changes in blood pressure, cardiac contractility, or heart rate.

This controlled not-randomized pilot study with repeated measures was conducted at the Touro University Nevada College of Osteopathic Medicine. Healthy 21-35 years old students and employees volunteered in the study. The experimental group received the three cranial osteopathic manipulative techniques, occipital-atlantal decompression, occipital-mastoid decompression, and compression of the fourth ventricle, consecutively applied. This study included two control groups; one group received sham manipulations, and the second group did not receive any manipulations and was the non-touch group.

The computerized MP150 BIOPAC System was used for data collection and analysis. The skin electrodes were used for the one-lead ECG and impedance cardiography. Digital data were recorded during the entire experimental protocol. The blood pressure was measured manually before and after the experimental procedure using blood pressure cuff and stethoscope. Cardiovascular responses to OMT were evaluated by using the heart rate variability test (HRV), calculating changes in cardiac contractility, and comparing changes in pre- and post- blood pressure readings.

An analysis of variance (ANOVA) with a Bonferroni post-hoc test was used to evaluate treatment effects. The type I error rate (alpha) was set at 0.05.

DETAILED DESCRIPTION:
Healthy, 21-35 year old, male and female volunteers were recruited from Touro University students, faculty and staff using a brochure, poster, e-mail or personal conversation. Each participant signed an informed consent form. Participants were allowed to participate in multiple experiments (in the experimental and control groups) at least 7 days after the last experiment.

Each subject's weight and height were measured before the procedure. Anthropometric measures were used in cardiac impedance analysis, and as descriptive statistics of the studied population. All cardiovascular parameters were recorded by using a non-invasive method. The disposable skin electrodes were used for impedance cardiography and a one-lead ECG.

The subjects were lying in the supine position and were asked to relax. All surface electrodes were connected to the computerized MP150 BIOPAC System for data recording. The duration of experimental protocol was about 30 minutes, and included three intervals: 10 minutes, pre-OMT rest phase (Rest); 8 to12 minutes (about 10 minutes) of the OMT/Sham (Manipulations); and 10 minutes post-OMT recovery phase (Recovery).

OMT and sham manipulations were administered by an osteopathic physician. The participants were told to lie supine with physician seated at the side of the table facing the participant. Cranial OMT included three techniques and was administered in the following sequence: occipital-atlantal decompression, occipital-mastoid joint, and compression of the fourth ventricle. Control subjects received the sham manipulative procedure or relaxed in supine position (non-touch control). The total duration of OMT controlled by an osteopathic physician and was about 10 minutes.

OMT and sham manipulations Occipital-atlantal decompression: Patient is in the supine position. The operator places the tip of a finger against the posterior tubercle of the atlas and holds that bone anteriorly, preventing it from moving posteriorly with the condyles as the patient nods or tips the head forward. This will release tension between the occipital condyles and the first cervical vertebrae.

Occipital-mastoid joint decompression: The occipital squama is gently moved forward and upward (anteriorly and superiorly) with the pads of the long finger, and the mastoid process of the temporal bone is lifted anterolaterally with the pads of the index fingers. This technique decompresses the jugular foramen, which the vagus nerve passes through.

Compression of the fourth ventricle: Manipulation is accomplished by having the operator's hands cupped to receive the lateral angles and supra-occiput on their thenar eminences. Gentle compression medially is maintained (generally 2 to 3 minutes) until tissue changes, such as a softening or increased motion, are noted in the supraoccipital area.

Sham: The osteopathic physician placed his hands on the skull of the subject and did not influence cranial motion. The sham manipulative procedure (SMP) was administered for 10 minutes.

All manipulations were administered by the osteopathic physician; experiments were conducted at Touro University Nevada. Data were collected by a non-invasive method using BIOPAC Systems, Inc. Equipment MP150 for data acquisition and analysis. The protocol consisted of three phases: rest before manipulations (10 min), manipulations (OMT) (approximately 10 min), and recovery after manipulations (10 min).

Data analysis Most cardiovascular response variables were measured at baseline, immediately after manipulation ("immediate response"), and at the end of protocol ("after rest"). The immediate responses and at the end of protocol were calculated on a percentage basis relative to baseline to control some individual variations.

The percent response variables were each analyzed in a three-way analysis of variance (ANOVA) which included time ("Immediate response", "after rest"), treatment (cranial manipulation, sham), and sex (male, female) as fixed effects. For significant interactions in the ANOVA, a Bonferroni post-hoc test was used to compare treatment effects within time, sex, or both. The type I error rate (alpha) was set at 0.05. The relationships among dependent variables were described with Spearman correlations between percent response variables within. Analyses were done in Rv3.5.1 (R Core Team 2018).

ELIGIBILITY:
Inclusion Criteria:

* Young adults

Exclusion Criteria:

* Clinical diagnosis of chronic cardiovascular diseases
* Clinical diagnosis of pulmonary diseases
* Clinical diagnosis of renal diseases
* Clinical diagnosis of diabetes mellitus
* Clinical diagnosis of endocrine disorders affecting the cardiovascular system
* Clinical diagnosis of pregnancy
* Clinical diagnosis of musculoskeletal conditions that can affect the use of the cranial OMTs
* Any acute illness that necessitates consulting a healthcare provider

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2013-10-04 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Change in heart rate variability immediately after manipulation | Baseline and 2 minutes after manipulation
  The heart rate variability test was used to study the effect of OMT on heart rate and, by inference, on autonomic nervous system activity. A decrease in heart rate accompanied by an increase in vagal and decrease in sympathetic activity would indicate parasympathetic activation by OMT.
Change in heart rate variability 10 min after manipulation | Baseline and 10 minutes after manipulation
  The heart rate variability test was used to study the effect of OMT on heart rate and, by inference, on autonomic nervous system activity. A decrease in heart rate accompanied by an increase in vagal and decrease in sympathetic activity would indicate parasympathetic activation by OMT.
Change in cardiac impedance immediately after manipulation | Baseline and 2 minutes after manipulation
  Changes in impedance cardiography were used to evaluate the effect of OMT on myocardial contractility.
Change in cardiac impedance 10 minutes after manipulation | Baseline and 10 minutes after manipulation
  Changes in impedance cardiography were used to evaluate the effect of OMT on myocardial contractility.
Change in blood pressure 10 minutes after manipulation | Baseline and 10 minutes after manipulation
  Blood pressure was measured by sphygmomanometer. Changes in blood pressure would indicate the effect of manipulation on vascular sympathetic tone.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Ioudina, MD, PhD, MS, Principal Investigator — Touro University Nevada

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: Starting 6 months after publication
Access Criteria: By direct contact with study authors

REFERENCES:
- [Background] Zurowska A, Malak R, Kolcz-Trzesicka A, Samborski W, Paprocka-Borowicz M. Compression of the Fourth Ventricle Using a Craniosacral Osteopathic Technique: A Systematic Review of the Clinical Evidence. Evid Based Complement Alternat Med. 2017;2017:2974962. doi: 10.1155/2017/2974962. Epub 2017 Oct 18. PMID 29234380
- [Background] Cardoso-de-Mello-E-Mello-Ribeiro AP, Rodriguez-Blanco C, Riquelme-Agullo I, Heredia-Rizo AM, Ricard F, Oliva-Pascual-Vaca A. Effects of the Fourth Ventricle Compression in the Regulation of the Autonomic Nervous System: A Randomized Control Trial. Evid Based Complement Alternat Med. 2015;2015:148285. doi: 10.1155/2015/148285. Epub 2015 Jun 14. PMID 26199632
- [Background] Cerritelli F, Carinci F, Pizzolorusso G, Turi P, Renzetti C, Pizzolorusso F, Orlando F, Cozzolino V, Barlafante G. Osteopathic manipulation as a complementary treatment for the prevention of cardiac complications: 12-Months follow-up of intima media and blood pressure on a cohort affected by hypertension. J Bodyw Mov Ther. 2011 Jan;15(1):68-74. doi: 10.1016/j.jbmt.2010.03.005. Epub 2010 May 8. PMID 21147421
- [Background] Cutler MJ, Holland BS, Stupski BA, Gamber RG, Smith ML. Cranial manipulation can alter sleep latency and sympathetic nerve activity in humans: a pilot study. J Altern Complement Med. 2005 Feb;11(1):103-8. doi: 10.1089/acm.2005.11.103. PMID 15750368
- [Background] Jakel A, von Hauenschild P. Therapeutic effects of cranial osteopathic manipulative medicine: a systematic review. J Am Osteopath Assoc. 2011 Dec;111(12):685-93. PMID 22182954

DOCUMENTS (1):
  • Study Protocol (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT05515926/Prot_000.pdf